CLINICAL TRIAL: NCT06180616
Title: Tirzepatide for the Treatment of Concurrent Type 1 Diabetes and Overweight or Obesity: A Placebo-Matched Randomised Controlled Trial
Brief Title: Tirzepatide for the Treatment of Concurrent Type 1 Diabetes and Overweight or Obesity
Acronym: TZP-T1D
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, Sarah Glastras, Associate Professor, Royal North Shore Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TZP-T1D
Record Dates: First submitted 2023-11-21; First posted 2023-12-22 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes Mellitus; Overweight and Obesity
Keywords: Tirzepatide; GLP-1/GIP Agonist
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Overweight; Obesity | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin Treatment (No Intervention): Participants will remain on their typical insulin therapy regime for 32 weeks
- Tirzepatide Treatment (Experimental): Participants will remain on their typical insulin therapy regime and will also receive tirzepatide (dose incremented to 15mg QW) for 32 weeks.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide will be self-administered subcutaneously by study participants via an injection. The drug will be taken weekly following the schedule: 4 weeks at 2.5 mg QW, 4 weeks at 5.0 mg QW, 4 weeks at 7.5 mg QW, 4 weeks at 10.0 mg QW, 4 weeks at 12.5 mg QW, 12 weeks at 15 mg QW.
  Modification of study drug will be performed if the participant is experiencing significant side effects and cannot tolerate the higher dosage of the study drug. In this instance, the study drug dosage will be reduced to the previously tolerated dosage and held at this dose for a further 4 weeks. One further attempt at dose escalation will be undertaken after 4 weeks, at the discretion of the participant and the study investigator. If recurrent side effects are experienced by the participant, the study drug will be returned to the previously tolerated dosage, and the prescription continued at this dosage for the remainder of the study.
  Arms: Tirzepatide Treatment

SUMMARY:
This study is a 2-arm, double blinded, randomised clinical trial where 40 participants will be assigned 1:1 to insulin treatment alone (control) or insulin treatment and tirzepatide treatment for 32 weeks. The primary objective is to demonstrate that tirzepatide treatment, dose incremented to 15mg QW for 32 weeks adjunctive to insulin treatment can reduce body weight in patients with T1D and overweight or obesity when compared to insulin treatment alone. The secondary objective is to demonstrate that tirzepatide treatment, dose incremented to 15mg QW for 32 weeks can improve glycaemic control (measured by hbA1c), improve time in range, reduce insulin requirements, and reduce the severity of comorbidities in people with obesity and T1D. This trial includes a 6 month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years at screening
* A clinical diagnosis of T1D for at least 12 months at time of screening
* Body mass index ≥ 27kg/m2
* HbA1c ≤ 10%
* Capable and willing to self-inject tirzepatide once per week
* In women of childbearing potential, a negative pregnancy test and willing to use effective contraception consistently for the duration of the study
* Able and willing to provide written informed consent for study participation
* Able and willing to use Easy Diet Diary
* Able and willing to keep an exercise log
* Willing to share devices data uploads
* Has current glucagon product to treat severe hypoglycaemia
* Has current ketone meters to check ketones

Exclusion Criteria:

* Age <18 years and >70 years
* A clinical diagnosis of diabetes type other than T1D
* HbA1c > 10%
* Use of GLP-1 receptor agonist within 1 month of study screening
* Use of any glucose lowering medications aside from insulin within 1 month of study screening
* History of hypersensitivity to investigational medicinal product or related product
* Obesity that is induced by other endocrine disorders
* Pregnancy or positive pregnancy test at time of screening, or unwilling to use effective contraception consistently for the duration of the study which is defined in Appendix 1
* Active proliferative diabetic retinopathy, maculopathy, or severe no proliferative diabetic retinopathy requiring acute treatment
* Known gastric emptying abnormality
* History of chronic or acute pancreatitis, uncontrolled hypertension, acute cardiovascular condition within 3 months
* No longer than 12 months of insulin treatment
* Not willing to use a NovoPen 6 to record insulin dosing if currently using multiple daily injections
* Insulin pump, CGM or smart phone devices are not compatible for data transfer
* Not willing to share device data
* Current use of any steroidal medication, or planned long-term steroidal treatment (>4 weeks) during the study period
* Serum triglycerides >500 mg/dL
* History of or plans for bariatric surgery during the study period
* eGFR <45 ml/min/1.73 m2
* History of severe hypoglycaemia (within 3 months of trial period)
* History of diabetic ketoacidosis (within 3 months of trial period)
* History of stroke (within 3 months of trial period)
* History of heart failure
* Planned coronary, carotid, or peripheral artery revascularisation
* History of acute or chronic liver disease
* History of allergy to any form of insulin, GLP-1RA or its excipients
* History of malignancy requiring chemotherapy, surgery, or radiation (within 5 years of trial period)
* History of multiple endocrine neoplasia type 2, familial thyroid cancer, or non-familial medullary thyroid cancer
* Presence or history of malignant neoplasms or in situ carcinomas (other than basal or squamous cell skin cancer, low-risk prostate cancer, or in situ carcinomas of the cervix or carcinoma in situ/high grade prostatic intraepithelial neoplasia) within 5 years before screening
* Have a pacemaker, or metal implants
* Participation in other intervention trials during the study period
* Existence of any additional health conditions or medical issues, including significant psychiatric disorders, that render a person unfit for the study at the discretion of the investigators

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Body weight | 32 weeks
  Percent body weight change (%)

SECONDARY OUTCOMES:
hbA1c | 32 weeks
  Change in hbA1c levels (%)
Time in range | 32 weeks
  Change in continuous glucose monitoring (CGM) metrics (time in range (3.9-10mmol/L))
Total daily insulin dose | 32 weeks
  Change in insulin dose (total daily dose, units/kg of body weight)
Insulin carbohydrate ratio | 32 weeks
  Change in insulin dose (insulin carbohydrate ratio (units per g))
Waist and neck circumference | 32 weeks
  Change in waist and neck circumference
Blood pressure | 32 weeks
  Change in blood pressure
Mean glucose | 32 weeks
  Change in continuous glucose monitoring (CGM) metrics (mean glucose)
Time in hypoglycaemia | 32 weeks
  Change in continuous glucose monitoring (CGM) metrics (time in hypoglycaemia (mild < 3.9, severe < 2.5mmol/L))
Time in hyperglycaemia | 32 weeks
  Change in continuous glucose monitoring (CGM) metrics (time in hyperglycaemia (mild >10, severe 13.9mmol/L))
Continuous glucose monitoring | 32 weeks
  Change in continuous glucose monitoring (CGM) metrics (SD)
Continuous glucose monitoring | 32 weeks
  Change in continuous glucose monitoring (CGM) metrics (CV)
Continuous glucose monitoring | 32 weeks
  Change in continuous glucose monitoring (CGM) metrics (CONGA)
Continuous glucose monitoring | 32 weeks
  Change in continuous glucose monitoring (CGM) metrics (J-index)
Continuous glucose monitoring | 32 weeks
  Change in continuous glucose monitoring (CGM) metrics (MAGE)
Total cholesterol | 32 weeks
  Change in lipid parameters (total cholesterol)
Triglyceride | 32 weeks
  Change in lipid parameters (triglyceride)
LDL-C | 32 weeks
  Change in lipid parameters (LDL-C)
HDL-C | 32 weeks
  Change in lipid parameters (HDL-C)
ACR | 32 weeks
  Change in albumin to creatinine ratio (ACR)
eGFR | 32 weeks
  Change in renal function (eGFR)
HSI | 32 weeks
  Change in NAFLD biomarker HSI. Hepatic steatosis defined as HSI > 36
FIB-4 | 32 weeks
  Change in NAFLD biomarker FIB-4. Hepatic steatosis defined as FIB-4 index ≥ 1.3 or < 1.3
Brachial-Ankle Pulse Wave Velocity using Ankle Brachial Index Machine | 32 weeks
  Change in Brachial-Ankle Pulse Wave Velocity (baPWV)
Arterial Stiffness using a Pulse Wave Tonometer | 32 weeks
  Change in arterial stiffness
Aortic Stiffness using a Pulse Wave Tonometer | 32 weeks
  Change in aortic stiffness
Left Ventricular Strain using Electrocardiogram | 32 weeks
  Change in left ventricular strain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data related to the primary and secondary outcomes may be shared upon reasonable request following publication. Data sharing will be considered for ethically approved research purposes and subject to data use agreements. IPD will not be shared if legal, ethical, or institutional constraints prevent it.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Purcell AR, Rodrigo N, Longfield MSG, Glastras SJ. Tirzepatide for the treatment of adults living with concurrent type 1 diabetes and overweight or obesity (TZP-T1D): a double-blind, placebo-matched randomised controlled trial protocol. BMJ Open. 2025 Sep 16;15(9):e093775. doi: 10.1136/bmjopen-2024-093775. PMID 40962353